CLINICAL TRIAL: NCT03978819
Title: Ability of the Analgesia Nociception Index Monitor to Distinguish Between Excessive Analgesia and Inadvertent Parasympathetic Nerve Stimulation During Surgery of Large Cerebellopontine Angle Tumours
Brief Title: ANI Parasympathetic Monitoring in Neurosurgery
Acronym: ANI
Status: Completed | Type: Observational
Sponsor: Association de Developpement de la Neuroanesthesie Reanimation (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Musa Sesay, Principal Investigator, Association de Developpement de la Neuroanesthesie Reanimation
Other Study IDs: DC 2015/143
Record Dates: First submitted 2019-05-21; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Bradycardia
Keywords: Analgesia nociception index; Parasympathetic nerve stimulation; Excessive analgesia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with large CPA tumors: Patients with large cerebellopontine angle tumors (>2 x 2cm) undergoing elective surgery
  Interventions: Device: ANI

INTERVENTIONS:
Device: ANI — ANI profiles during IPNS (bradycardia/asystole) or excessive analgesia.
  During surgery continuous monitoring of ANI, HR and Remifentanil effect site concentration was done and recorded. Event markers were placed at the onset of bradycardia, asystole and the coincidence of ANI>80 + Remifentanil >6ng/mL). ANI values of 1 min before and 1 min after the event were used for analysis.

SUMMARY:
Surgery of large cerebellopontine angle (CPA) tumors (>2 x 2 cm diameter), with compression of the pons exposes the patient to inadvertent parasympathetic nerve stimulation (IPNS) leading to bradycardia and asystole.

The analgesia nociception index (ANI) monitor assesses the balance between analgesia and nociception through the detection of parasympathetic tone. ANI >80 generally denotes excessive analgesia (EA). The main objective of this study was to determine whether ANI values for IPNS are different or the same as ANI values for EA. This study also aims at calculating the number of patients with IPNS and EA during surgery of large CPA tumours.

DETAILED DESCRIPTION:
Bradycardia and asystole are potential life threatning complications during surgery of large cerebellopontine angle (CPA) tumors (>2 x 2 cm diameter), with compression of the pons.The incidence of such complications are unknown. One of the plausible mechanisms is inadvertent parasympathetic nerve stimulation (IPNS) due to the proximity of this cranial nerve to the CPA tumor. Monitoring parasympathetic nerve activity may provide further insight to the implication of this cranial nerve in the cardiac complications observed during surgery of large CPA tumors. The analgesia nociception index (ANI) monitor assesses the balance between analgesia and nociception through the detection of parasympathetic tone. Despite the abundant clinical reports about this index, to the knowledge of the investigators, only a few studies have been published in the neurological setting. Moreover, there are no data reporting the parasympathetic profile (measured by the ANI monitor) in situations of IPNS and EA. Are these profiles the same or different? Such is the main question this study thrives to answer. Understanding the behavior of parasympathetic nerve activity in this context could help provide the appropriate management strategy.

In order to answer this question, participants undergoing elective large CPA tumor surgery were included in this prospective observational study. Standard cardiorespiratory monitoring including heart rate (HR) was done. Target-controlled anesthesia with Propofol and Remifentanil was guided by a bispectral index of 30-40 and an ANI of 50-70 respectively. Data was continuously recorded with event markers at the onset of bradycardia (HR < 45 bpm), asystole and the coincidence of ANI > 80 with Remifentanil site effect > 6 ng.ml-1 (defined as excessive analgesia).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective surgery of large cerebellopontine angle tumors

Exclusion Criteria:

* age below 18yr
* arrhythmia
* preoperative use of vagolytics, β-blockers and clonidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female with large cerebellopontine angle tumors (>2 x 2 cm)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Differences in instantaneous ANI (ANIi) values during bradycardia versus ANIi values when Remifentanil effect size concentration >6ng/mL | ANIi values recorded at Day 1 only during surgery (duration: 4-6 hours)
  ANI, HR and Remifentanil effect site concentration were continuously recorded with event markers on the ANI monitor at the onset of bradycardia (HR<45 bpm) or Remifentanil effect site concentration>6ng/mL
Differences in the area under the ROC curves between ANI values for IPNS and EA analgesia | ANIi values recorded at Day 1 only during surgery (duration: 4-6 hours)
  ROC curves were built at different ANIi for IPNS or EA

SECONDARY OUTCOMES:
Percentages of IPNS and EA cases | Cases observed at Day 1 only during surgery (duration: 4-6 hours)
  The percentages of IPNS or EA cases on the overall study population were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Sesay, M.D, Principal Investigator — ADNR, Neuroanesthesia and Critical Care, 33076 Bordeaux, France; Matthieu Biais, M.D., PhD, Study Director — Neuroanesthesia and Critical Care, CHU University Bordeaux; Karine Nouette-Gaulain, M.D., Ph.D, Study Chair — Neuroanesthesia and Critical Care, CHU University Bordeaux
Locations (1):
- CHU Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renowden S. Imaging of the cerebello-pontine angle. Pract Neurol. 2014 Oct;14(5):e2. doi: 10.1136/practneurol-2014-000949. Epub 2014 Aug 12. No abstract available. PMID 25118279
- [Background] Sesay M, Vignes JR, Stockle M, Mehsen M, Boulard G, Maurette P. [Spectral analysis of the ECG R-R interval permits early detection of vagal responses to neurosurgical stimuli]. Ann Fr Anesth Reanim. 2003 May;22(5):421-4. doi: 10.1016/s0750-7658(03)00094-7. French. PMID 12831969
- [Background] De Jonckheere J, Rommel D, Nandrino JL, Jeanne M, Logier R. Heart rate variability analysis as an index of emotion regulation processes: interest of the Analgesia Nociception Index (ANI). Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:3432-5. doi: 10.1109/EMBC.2012.6346703. PMID 23366664
- [Background] Jeanne M, Clement C, De Jonckheere J, Logier R, Tavernier B. Variations of the analgesia nociception index during general anaesthesia for laparoscopic abdominal surgery. J Clin Monit Comput. 2012 Aug;26(4):289-94. doi: 10.1007/s10877-012-9354-0. Epub 2012 Mar 28. PMID 22454275
- [Background] Robin F, Sesay M, Kolanek B, Pena D, Penna M, Morel-Locket L et al. The analgesia nociception index monitor (ANI) can detect indvertent vagal stimulation during surgery of cerebello-pontine angle tumors. Br J Anaesth 2013;111: https: // doi.org/10.1093/bja/el_10195
- [Background] Kommula LK, Bansal S, Umamaheswara Rao GS. Analgesia Nociception Index Monitoring During Supratentorial Craniotomy. J Neurosurg Anesthesiol. 2019 Jan;31(1):57-61. doi: 10.1097/ANA.0000000000000464. PMID 28991059
- [Background] Theerth KA, Sriganesh K, Reddy KM, Chakrabarti D, Umamaheswara Rao GS. Analgesia Nociception Index-guided intraoperative fentanyl consumption and postoperative analgesia in patients receiving scalp block versus incision-site infiltration for craniotomy. Minerva Anestesiol. 2018 Dec;84(12):1361-1368. doi: 10.23736/S0375-9393.18.12837-9. Epub 2018 Jul 9. PMID 29991223
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Galley HF. Editorial II: Solid as a ROC. Br J Anaesth. 2004 Nov;93(5):623-6. doi: 10.1093/bja/aeh247. No abstract available. PMID 15472141

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03978819/Prot_SAP_000.pdf